CLINICAL TRIAL: NCT02953184
Title: Marched Pair Study of the Standard Chemotherapy 4doxorubicin Plus Cyclophosphamide(AC) 60 + 4 Docetaxel Protocol Versus 4 PLD C35+4 Docetaxel in Neoadjuvant Chemotherapy of Breast Cancer
Brief Title: Marched Pair Study Conventional Doxorubicin(DOX) Versus Pegylated Liposomal Doxorubicin(PLD) Neoadjuvant Chemotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jilin University (Other)
Responsible Party: Principal Investigator, Aiping shi, Professor, Jilin University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016yx238
Record Dates: First submitted 2016-10-08; First posted 2016-11-02 (Estimated); Last update posted 2017-12-29 (Actual); Status verified 2017-12

CONDITIONS: Antineoplastic Combined Chemotherapy Protocols
Keywords: neoadjuvant chemotherapy; Pegylated liposomal doxorubicin; breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — liposomal doxorubicin; Cyclophosphamide; Docetaxel; Dexrazoxane; Folic Acid; Doxorubicin; pirarubicin; Injections; Mastectomy, Segmental; Mastectomy, Modified Radical; Mastectomy; Sentinel Lymph Node Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- conventional Doxorubicin plus C-T (Active Comparator): AC-T regimen 8 cycles ,60mg/M2 conventional Doxorubicin will be used as active comparator. four cycles of Doxorubicin plus 600mg/m2 Cyclophosphamide every three weeks followed 4 cycles of 100mg/m2 Taxotere, every three weeks for one cycle.Dexrazoxane (DZR)will be used for protecting cardiac toxicity.Patients will undergo Modified Radical Mastectomy or Breast Conserved Surgery or Axillary Lymph Node Dissection(ALND) or Sentinel Lymph Node Biopsy（SLNB） after 8 cycles of chemotherapy
  Interventions: Drug: Cyclophosphamide; Drug: Taxotere; Drug: Dexrazoxane (DZR); Drug: Doxorubicin; Procedure: Breast Conserved Surgery; Procedure: Modified Radical Mastectomy; Procedure: Sentinel Lymph Node Biopsy（SLNB）
- PLD plus C -T (Experimental): Pegylated Liposomal Doxorubicin(PLD) plus Cyclophosphamide followed Taxotere 8 cycles.35mg/M2 PLD will be used as experimental medicine. four cycles of PLD plus 600mg/m2 Cyclophosphamide every three weeks followed 4 cycles of 100mg/m2 Taxotere , every three weeks for one cycle.Vitamin B will be used for protecting hand-foot syndrome(HFS).Patients will undergo Modified Radical Mastectomy or Breast Conserved Surgery or Axillary Lymph Node Dissection(ALND) or Sentinel Lymph Node Biopsy（SLNB） after 8 cycles of chemotherapy
  Interventions: Drug: Pegylated Liposomal Doxorubicin; Drug: Cyclophosphamide; Drug: Taxotere; Drug: vitamin B; Procedure: Breast Conserved Surgery; Procedure: Modified Radical Mastectomy; Procedure: Sentinel Lymph Node Biopsy（SLNB）

INTERVENTIONS:
Drug: Pegylated Liposomal Doxorubicin — 35mg/m2 iv drop during the first 4 cycles every three week
  Other Names: liposome doxorubicin injection
  Arms: PLD plus C -T
Drug: Cyclophosphamide — 600mg/m2 IV drop during the first 4 cycles every three week
  Other Names: cytoxan
Drug: Taxotere — 100mg/m2 IV drop during the last 4 cycles every three week
  Other Names: Docetaxel
Drug: Dexrazoxane (DZR) — DZR will be administrated for protecting Cardiac toxicity in the group of Active comparator.
  Other Names: DZR
  Arms: conventional Doxorubicin plus C-T
Drug: vitamin B — Vitamin B will be administrated for protecting HFS in PLD group
  Other Names: Compound Vitamin B
  Arms: PLD plus C -T
Drug: Doxorubicin — 60mg/m2 Doxorubicin IV drop during the first 4 cycles every three week
  Other Names: Pirarubicin Hydrochloride for injection
  Arms: conventional Doxorubicin plus C-T
Procedure: Breast Conserved Surgery — Patients will undergo Breast Conserved Surgery if the tumor/breast ratio is proper and she demands to conserve the breast after 8 cycles of chemotherapy
  Other Names: segmental mastectomy and ALND
Procedure: Modified Radical Mastectomy — Patients will undergo Modified Radical Mastectomy if she does not keep her breast after 8 cycles of chemotherapy
  Other Names: Mastectomy and ALND
Procedure: Sentinel Lymph Node Biopsy（SLNB） — Patients will undergo Sentinel Lymph Node Biopsy（SLNB） if the evaluation of lymph node are negative after 8 cycles of chemotherapy
  Other Names: Sentinel Lymph Node(SLN)

SUMMARY:
The regimen PLD plus cyclophosphamide 4 cycles followed by paclitaxel or docetaxel 4 cycles(noted in phase II CAPRICE) will be used as experimental group. The regimen will be compared to the standard treatment of doxorubicin plus cyclophosphamide(AC) 4 cycles followed by paclitaxel or docetaxel 4 cycles[noted in National Comprehensive Cancer Network (NCCN) guideline].

DETAILED DESCRIPTION:
Purpose :Anthracycline based chemotherapy regimen is the milestone on the treatment of breast cancer . A sequential protocol, using docetaxel or Paclitaxel after an anthracycline-based combination is primary treatment for high-risk breast cancer .Despite its efficient antitumor activity profile, the use of conventional anthracycline in clinical practice is limited due to it's the risk of cardiac toxicity. The meta analysis show that subclinical cardiotoxicity was 17.9% whereas the incidence of clinically overt cardiotoxicity was 6.3%. Overall cardiovascular events occurred in 10.6%(Lotrisone , Am J Cardiol. 2013).Many patients have healed from breast cancer while they are snatched lives because of heart issue from chemotherapy using anthracycline. There are a lot of clinical trials exploring the possibilities of chemotherapy regimen without anthracycline ,however the recent result has shown anthracycline is indispensible for the patients whose axillary nodes are involved or triple negative breast cancer (ASCO 2016 ).So our target is to find a kind of anthracycline which is of equal efficiency with conventional anthracycline while less cardiac toxicity. Pegylated Liposomal Doxorubicin(PLD) is a novel kind of anthracycline. It distributes into cardiac cells lowly and releases Doxorubicin (DOX) slower to avoid peak plasma concentration, so it is of significant less cardiotoxicity compared to free DOX. It also achieve non-inferior efficacy at 50mg/m2 to conventional anthracycline in Metastatic Breast Cancer (MBC).( M. E. R. O'Brien, ,Annals of Oncology,2004;).

PLD 35mg/m2 in combination with paclitaxel showed an overall response rate of 71% ,tolerating toxicity of the skin(3% hand-foot syndrome)and rare cardiac event( H. Gogas1, Annals of Oncology, 2002;Gil-Gil , Breast Cancer Res Treat. 2015)However, There are a crucial question is to know if 35mg/m2 PLD has equivalent efficacy with less cardiac toxicity compared with 60 mg/m2 DOX in adjuvant chemotherapy for all patients.

The regimen PLD plus cyclophosphamide 4 cycles followed by paclitaxel or docetaxel 4 cycles(noted in phase II CAPRICE)will be used as experimental group. The regimen will be compared to the standard treatment of doxorubicin plus cyclophosphamide (AC)4 cycles followed by paclitaxel or docetaxel 4 cycles(noted in NCCN guideline).

Condition Intervention Phase

Individualized Chemotherapy Drug: Pegylated Liposomal Doxorubicin(PLD) Drug: Doxorubicin(DOX)

Drug: Cyclophosphamide Drug: docetaxel or Paclitaxel Phase 2

Study Type: Interventional Study Design: Allocation: assignment based on patients desire Endpoint Classification: Safety/Efficacy Study Intervention Model: Marched pair Parallel Assignment Masking: Open Label Primary Purpose: Treatment

ELIGIBILITY:
Inclusion Criteria:

* Patient with histological proof of invasive cancer, whose clinical tumor diameter is > 2 cm, or < 2 cm, but Axillary lymphnodes are involved .There is no metastatic Imaging findings.
* Stage II,III tumor, non-metastatic, grade II - III
* Performance Status = 0-1 World Health Organization (WHO).
* Patient non pretreated for breast cancer.
* Patient without cardiac pathology and without anthracyclines contra-indication (assessed by normal ejection fraction).
* Normal haematological, renal and hepatic functions : platelets > 100. 109 /l, Hb > 10 g/dl, normal bilirubin serum , Aspartate transaminase(ASAT) and Alanine Aminotransferase(ALAT) < 2,5 Upper Limit of Normal (ULN), alkaline phosphatases < 2,5 ULN, creatinin < 140 µmol/l or creatinin clearance > 60 ml/min
* Written informed consent dated and signed by the patient

Exclusion Criteria:

* All other breast cancers than those described in inclusion criteria, in particular inflammatory and/or neglected (T4b or T4d) forms.
* Patient presenting with intraduct cancer in situ.(DCIS)
* Grade I well differentiated tumor.
* Non measurable lesion, in the two diameters, whatever radiological methods used.
* Patient already operated for breast cancer or having had primary axillar node dissection.
* Patient presenting with cancer in other system.
* Any psychological, familial, sociological or geographical condition that may potentially hamper compliance with the study protocol and follow up schedule, assessed with the patient prior to registration in the trial

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2016-11; Primary Completion 2019-11 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
improvement of pathological complete response（PCR) | at th 26th weeks of treatment since recruitment (after 8 cycles of neoadjuvant chemotherapy when the patient will undergo surgery)
  Pathological evaluation after sugary

SECONDARY OUTCOMES:
Tolerance according to Common Terminology Criteria Adverse Events (CTCAE) Version 4.0 | at 3rd ,6th,9th,12th, 15 ,18,21,24th weeks since recruitment (after each cycle of chemotherapy) ; half year ,1 year , one and half year ,two years since recruitment
  Cardiogram Cardiac sonography, examination of Cardiac Marker if necessary and Questionaire Survey about Side Effect
Clinical Response Rate | at 3rd ,6th,9th,12th, 15 ,18,21,24th weeks since recruitment （after each cycle of chemotherapy）
  ultrasound of breast and Pathological reports

CONTACTS AND LOCATIONS:
Overall Officials: Aiping Shi, Doctor, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: Jan 1,2018 to Dec ,31,2020

REFERENCES:
- [Background] Early Breast Cancer Trialists' Collaborative Group (EBCTCG); Peto R, Davies C, Godwin J, Gray R, Pan HC, Clarke M, Cutter D, Darby S, McGale P, Taylor C, Wang YC, Bergh J, Di Leo A, Albain K, Swain S, Piccart M, Pritchard K. Comparisons between different polychemotherapy regimens for early breast cancer: meta-analyses of long-term outcome among 100,000 women in 123 randomised trials. Lancet. 2012 Feb 4;379(9814):432-44. doi: 10.1016/S0140-6736(11)61625-5. Epub 2011 Dec 5. PMID 22152853
- [Background] Lotrionte M, Biondi-Zoccai G, Abbate A, Lanzetta G, D'Ascenzo F, Malavasi V, Peruzzi M, Frati G, Palazzoni G. Review and meta-analysis of incidence and clinical predictors of anthracycline cardiotoxicity. Am J Cardiol. 2013 Dec 15;112(12):1980-4. doi: 10.1016/j.amjcard.2013.08.026. Epub 2013 Sep 25. PMID 24075281
- [Background] Jones S, Holmes FA, O'Shaughnessy J, Blum JL, Vukelja SJ, McIntyre KJ, Pippen JE, Bordelon JH, Kirby RL, Sandbach J, Hyman WJ, Richards DA, Mennel RG, Boehm KA, Meyer WG, Asmar L, Mackey D, Riedel S, Muss H, Savin MA. Docetaxel With Cyclophosphamide Is Associated With an Overall Survival Benefit Compared With Doxorubicin and Cyclophosphamide: 7-Year Follow-Up of US Oncology Research Trial 9735. J Clin Oncol. 2009 Mar 10;27(8):1177-83. doi: 10.1200/JCO.2008.18.4028. Epub 2009 Feb 9. PMID 19204201
- [Background] Gogas H, Papadimitriou C, Kalofonos HP, Bafaloukos D, Fountzilas G, Tsavdaridis D, Anagnostopoulos A, Onyenadum A, Papakostas P, Economopoulos T, Christodoulou C, Kosmidis P, Markopoulos C. Neoadjuvant chemotherapy with a combination of pegylated liposomal doxorubicin (Caelyx) and paclitaxel in locally advanced breast cancer: a phase II study by the Hellenic Cooperative Oncology Group. Ann Oncol. 2002 Nov;13(11):1737-42. doi: 10.1093/annonc/mdf284. PMID 12419745
- [Background] Gil-Gil MJ, Bellet M, Morales S, Ojeda B, Manso L, Mesia C, Garcia-Martinez E, Martinez-Janez N, Mele M, Llombart A, Pernas S, Villagrasa P, Blasco C, Baselga J. Pegylated liposomal doxorubicin plus cyclophosphamide followed by paclitaxel as primary chemotherapy in elderly or cardiotoxicity-prone patients with high-risk breast cancer: results of the phase II CAPRICE study. Breast Cancer Res Treat. 2015 Jun;151(3):597-606. doi: 10.1007/s10549-015-3415-2. Epub 2015 May 16. PMID 25981896
- [Background] O'Brien ME, Wigler N, Inbar M, Rosso R, Grischke E, Santoro A, Catane R, Kieback DG, Tomczak P, Ackland SP, Orlandi F, Mellars L, Alland L, Tendler C; CAELYX Breast Cancer Study Group. Reduced cardiotoxicity and comparable efficacy in a phase III trial of pegylated liposomal doxorubicin HCl (CAELYX/Doxil) versus conventional doxorubicin for first-line treatment of metastatic breast cancer. Ann Oncol. 2004 Mar;15(3):440-9. doi: 10.1093/annonc/mdh097. PMID 14998846

DOCUMENTS (1):
  • Informed Consent Form (2016-10-08): https://cdn.clinicaltrials.gov/large-docs/84/NCT02953184/ICF_000.pdf